CLINICAL TRIAL: NCT05072054
Title: Comparison of Effects of Atorvastatin Versus Rosuvastatin Treatment on Cardiac Function and Inflammation in Patients With Chronic Heart Failure With Reduced Ejection Fraction: A Randomised, Double Blind Clinical Study
Brief Title: Comparison of Effects of Atorvastatin Versus Rosuvastatin on Cardiac Function in Heart Failure Patients
Acronym: ASTRO-CHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Indian Council of Medical Research (Other Government)
Responsible Party: Principal Investigator, Ashish Kakkar, Associate Professor, Department of Pharmacology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PGIMER-CV-2019
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Atorvastatin; Rosuvastatin; Heart failure
MeSH Terms: conditions — Heart Failure | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind clinical study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized to two arms in ratio 1:1 using computer-generated random list. Patients, investigator and care provider will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin arm (Experimental): Tablet Atorvastatin 40mg once daily at bed-time given for 6 months
  Interventions: Drug: Atorvastatin Oral Tablet
- Rosuvastatin arm (Active Comparator): Tablet Rosuvastatin 20mg once daily at bed-time given for 6 months
  Interventions: Drug: Rosuvastatin Oral Tablet

INTERVENTIONS:
Drug: Atorvastatin Oral Tablet — Atorvastatin 40 mg
  Arms: Atorvastatin arm
Drug: Rosuvastatin Oral Tablet — Rosuvastatin 20 mg
  Arms: Rosuvastatin arm

SUMMARY:
Statins have a protective effect in patients with established heart failure because of their lipid-lowering and pleiotropic effects. There is no randomized controlled trial comparing lipophilic versus hydrophilic statins in these patients (head to head comparison). The best evidence so far is from a meta-analysis in which the authors did an adjusted indirect comparison between lipophilic statins and rosuvastatin and found that lipophilic statins were associated with significantly lower incidence of all-cause mortality, cardiovascular mortality, and hospitalization for worsening heart failure compared to rosuvastatin (hydrophilic statin) among patients with heart failure. So, the investigators plan to conduct a randomized controlled trial comparing the effects of atorvastatin and rosuvastatin on cardiac function in patients with heart failure with reduced ejection fraction.

DETAILED DESCRIPTION:
HMG CoA reductase inhibitors or Statins have been widely used for primary prevention and secondary prevention of atherosclerotic cardiovascular disease. Also, the protective effect of statins has been observed in patients with established heart failure because of their lipid-lowering and pleiotropic effects.

Various randomized and non-randomized clinical trials have evaluated statins like Atorvastatin, Rosuvastatin, Simvastatin, Pitavastatin and reported improved clinical outcomes in patients with heart failure with reduced ejection fraction as well as heart failure with preserved ejection fraction. Similar benefits on improved cardiac function, reduced inflammation, and improved mortality have been seen in small randomized controlled trials (RCTs) with Atorvastatin. The two large RCTs - Controlled Rosuvastatin Multinational Study in Heart Failure (CORONA) and Gruppo Italiano per lo Studio della Sopravvivenza nell'Insufficienza cardiac (GISSI-HF) - which compared Rosuvastatin versus placebo, failed to show statistically significant benefits in mortality outcomes in heart failure patients compared to placebo, although CORONA trial did show a significant reduction in hospital admissions but not on mortality.

However, these two large trials only compared one statin i.e rosuvastatin versus placebo; which is a hydrophilic statin. Statin is not a uniform class of drugs. They differ in their pleiotropic effects based on lipophilic nature. There is evidence that lipophilic statins enter cells via passive diffusion and are widely distributed to various tissues including cardiac tissues where it exerts pleiotropic actions whereas uptake of hydrophilic statins is via carrier-mediated mechanisms and is restricted to the liver, thus reduced the capacity of non-lipid effects on extra-hepatic tissues.

Currently, there is no RCT comparing lipophilic statin versus hydrophilic statin (head to head comparison). The best evidence so far is from a meta-analysis which is an adjusted indirect comparison between lipophilic statins and rosuvastatin. They found that lipophilic statins were associated with a significantly lower incidence of all-cause mortality, cardiovascular mortality, and hospitalization for worsening heart failure compared to rosuvastatin (hydrophilic statin) among patients with heart failure. So, the investigators plan to conduct a randomized controlled trial comparing the effects of atorvastatin and rosuvastatin on cardiac function and inflammation in patients with heart failure with reduced ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender,18-65 years of age
2. Left ventricular ejection fraction <40% as assessed by 2D echocardiography
3. NYHA class II-III
4. CHF patients currently optimized on standard treatment for at least 1 month before enrolment and on an OPD basis treatment
5. Ready to give written informed consent
6. Willing to comply with the study protocol

Exclusion Criteria:

1. Known hypersensitivity to statins
2. NYHA class IV patient
3. Serum creatinine >3 mg/dl
4. Significant liver disease: SGOT/SGPT >3 times the upper limit of normal (ULN) or >2.5 times the ULN in symptomatic patients
5. Patient on an enzyme inducer or inhibitor currently
6. Any malignancy or patient on chemotherapeutic agents
7. Pregnant or lactating females
8. Patients who have participated in another trial within the past 3 months
9. Patient with uncontrolled diabetes mellitus (HbA1c >7 g%)/ uncontrolled hypertension (BP >140/90 mmHg despite in ≥3 antihypertensive drugs)
10. Patient with HIV/ HBV / HCV infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-16 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
To compare the effect of atorvastatin and rosuvastatin on LVEF | Measurements at enrolment (baseline), 3 month and 6 months
  Change from baseline in Left ventricular ejection fraction (LVEF) measured by 2D Echocardiography after atorvastatin or rosuvastatin treatment
To compare the effect of atorvastatin and rosuvastatin on NT-ProBNP | Measurements at enrolment (baseline), 3 months and 6 months
  Change from baseline in NT-ProBNP (cardiac marker) after atorvastatin or rosuvastatin treatment.

SECONDARY OUTCOMES:
To compare the effect of atorvastatin and rosuvastatin on IL-6 | Measurements at enrolment (baseline) and 6 months
  Change from baseline in IL-6 levels after atorvastatin or rosuvastatin treatment
To compare the effect of atorvastatin and rosuvastatin on hsCRP | Measurements at enrolment (baseline), 3 month and 6 months
  Change from baseline in hsCRP levels after atorvastatin or rosuvastatin treatment.
To compare the effect of atorvastatin and rosuvastatin on Minnesota living with heart failure questionnaire (MLHFQ) | Measurements at enrolment (baseline), 3 month and 6 months
  Change from baseline in Minnesota living with heart failure questionnaire (MLHFQ) after atorvastatin or rosuvastatin treatment. MLHFQ consists of 21 questions and each question has a score from 0 to 5.
  The total score ranges from 0 to 105, with higher scores indicating greater impairment in health related quality of life.
To compare the effect of atorvastatin and rosuvastatin on 6-minute walk test (6MWT) | Measurements at enrolment (baseline), 3 month and 6 months
  Change from baseline in 6-minute walk test (6MWT) after atorvastatin or rosuvastatin treatment.
Compare incidence of hospitalization for worsening of heart failure at 6 months in atorvastatin and rosuvastatin group | Analysis at 6 months
  Incidence of hospitalization due to worsening of heart failure in 6 months in both groups
Compare incidence of adverse events and major adverse events including all-cause mortality, non-fatal MI, stroke in atorvastatin and rosuvastatin group. | Analysis at 6 months
  Incidence of adverse events including serious adverse events in 6 months in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ashish K Kakkar, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No